CLINICAL TRIAL: NCT06226298
Title: Benefits of the Xiaxi Postural Hammock and a Xiaxi Exercise Program: A Randomized Controlled Trial
Brief Title: Benefits of the Xiaxi Postural Hammock and a Xiaxi Exercise Program
Acronym: XHEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAM_23
Record Dates: First submitted 2023-11-07; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Low Back Pain; Exercise
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiaxi (Experimental): The experimental group will lie in the Xiaxi postural hammock for 10 minutes for 5 days.
  Interventions: Device: Xiaxi postural hammock
- Control (Active Comparator): The control group will lie on a mat on the floor for 10 minutes, 5 days of intervention.
  Interventions: Behavioral: Yoga mat

INTERVENTIONS:
Device: Xiaxi postural hammock — Lie in the Xiaxi postural hammock for 10 minutes for 5 days.
  Arms: Xiaxi
Behavioral: Yoga mat — Lie in the Yoga mat for 10 minutes for 5 days.
  Arms: Control

SUMMARY:
Chronic low back pain is one of the main causes of pain, dysfunction and disability worldwide. In Spain, 93% of the population has had back pain in the last year, and it is estimated that 50% of sick leave is due to this cause. This entails a great socioeconomic burden, since it is the main cause of absenteeism from work and the excessive use of therapeutic services.

Musculoskeletal disorders are related and associated with psychologically stressful jobs, that is, with psychosocial factors at work and related work stressors, such as time pressure, low job control, poor social or supervisor support, effort-reward imbalance or work-life conflict. Clinical management of both situations encompasses a variety of approaches, including medication and early physical exercise, which have shown promise in reducing pain and improving function.

A novel approach to address these problems is the use of Xiaxi, a patented postural hammock with multiple angles of inclination that promotes relaxation and elongation of the posterior chain, thereby improving overall well-being. Combining the use of Xiaxi with a comprehensive program of strengthening, stretching and relaxation exercises could offer benefits in the prevention and reduction of back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Presence of back pain.

Exclusion Criteria:

* Have undergone surgery of the spine, ischiosural muscles, psoas-iliac, pectoral and rotator cuff.

  * to have any structured spinal spine alteration diagnosed by health personnel.
  * have had a rupture of the ischiosural, psoas-iliac, pectoral and rotator cuff muscles in the last year or during the intervention.
  * have any type of injury that prevents you from performing the initial assessment in the first week of the procedure.
  * to have practiced vigorous physical exercise on the day of the investigation or 24 hours before the initial or final assessment.
  * having eaten large meals on the days of the investigation
  * less than two hours had elapsed since any prolonged recumbent rest at the start of the assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for pain | 1 minute
  The VAS will be used to assess the level of pain intensity. The VAS scale allows measuring the intensity of pain described by the patient with maximum reproducibility between observers. It consists of a horizontal line of 10 centimeters, at the ends of which are the extreme expressions of a symptom. On the left side is located the absence or lower intensity and on the right side the higher intensity. The patient is asked to mark on the line the point indicating the intensity and it is measured with a millimeter ruler. The intensity is expressed in centimeters or millimeters. It is a common, simple, well constructed, validated and reliable method.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) for Physical Activity | 5 minutes
  The IPAQ is a questionnaire with internationally accepted validity and reliability, which allows measuring the degree of activity in different populations between 15 and 69 years of age. This questionnaire asks about physical activity related to work, transportation, home activity, leisure time and determines the degree of physical activity according to the metabolic equivalents consumed during such activity.
General health status, the "SF-36", for quality of life | 5 minutes
  For the assessment of general health status, the "SF-36" health status questionnaire will be used. The SF-36 health questionnaire is a widely used outcome instrument to assess health-related quality of life. It is a generic multidimensional instrument validated for several pathologies. The physical component summary of the SF36 assesses functional capacity, physical aspects, pain and general health, while its mental component summary assesses vitality, social functioning, emotional aspects and mental health.
Satisfaction With Life Scale (SWLS) questionnaire, for quality of life | 5 minutes
  The SWLS is a useful instrument for academic research in social, medical and other disciplines, as it has demonstrated a high degree of reliability in several studies, appropriate internal consistency among items, correlations between items and adequate validity. The instrument consists of a brief 5-question questionnaire designed to evaluate people's general satisfaction with their lives. It requires approximately one to five minutes of the respondent's time to complete. Responses are recorded on a 7-point Likert rating scale, where 1 represents "strongly disagree" and 7 means "strongly agree". Scores obtained can range from 5 to 35, with higher scores indicating that the person perceives that important areas of his or her life are going well, while lower scores indicate the opposite.
Perceived Stress Scale (PSS), for stress | 5 minutes
  The PSS is a scale designed to measure the degree to which individuals rate situations in their lives as stressful. The items assess the degree to which people consider life to be unpredictable, uncontrollable, or overloaded, central components of stress. The scale includes questions designed to assess the current level of stress experienced by the subject. It is a brief scale, consisting of only 14 items, takes only a few minutes to administer, and is easily scored.
The Hospital Anxiety and Depression Scale (HADS), for Anxiety and Depression | 5 minutes
  The HADS will be used to assess anxiety and depression symptoms. The HADS is a brief two-dimensional self-completed questionnaire designed to assess anxiety and depression symptoms in individuals with physical health problems. It consists of 14 items, 7 of which focus on anxiety symptoms and the other 7 on depressive symptoms. The HADS is considered a valuable tool for screening for these psychological problems in medical settings because of its brevity, ease of administration, and good psychometric properties.
Oswestry Low Back Pain Disability Scale, for disability | 5 minutes
  The Oswestry Low Back Pain Disability Scale will be used to assess the level of disability due to pain. This scale is the most widely used, together with the Roland-Morris scale, in the evaluation of the patient with low back pain to measure its functional repercussion on activities of daily living. It is made up of ten items related to activities of daily living. For each item there are 6 possible answers ranging from no disability [0] to total disability [5]. The Spanish version, which has been translated and culturally adapted, was used.
Pressure pain threshold (PPT), for pain | 5 minutes
  A digital algometer (Model FXD 10, Wagner Instruments, Greewich, CT, USA) that measures pressure in kg/cm2 will be used to assess the PPT. The UDP is defined as the minimum pressure necessary for the pressure sensation to begin to be perceived as painful. To assess it, increasing pressure is applied to the upper portion of the trapezius muscle on the right side at a rate of one kilogram per second until the subject indicates that the sensation begins to be painful. The study subject was in a seated position. To improve accuracy, the investigator in charge of taking this measurement precisely marked the area where the measurement would be taken with a marker. Each measurement would be taken three times and the arithmetic mean was taken to establish the final value collected. Subsequently, it was evaluated in the left upper trapezius muscle, in the right quadratus lumborum muscle and in the left quadratus lumborum muscle, following the procedure previously described.
Angular and a linear test for the assessment of hamstring extensibility for flexibility | 2 minutes
  For the assessment of hamstring extensibility, angular tests and a linear test will be performed. As a reference angular test, the straight leg raising test will be performed, assessing both legs passively (EPRPassive) and actively (EPRActive). The measurement will be performed with an inclinometer (Baseline, model Bubble ® inclinometer, White Plains, NY 10602 (USA). The sit-and-reach test will also be performed, assessing both the pelvic tilt (with the inclinometer) and the distance reached in the test (linear measurement). The tests will be performed in a randomized order and by the same investigator for each test.
Modified-Modified Schober Test, for flexibility | 2 minutes
  For the assessment of lumbar spine flexibility, the Modified-Modified Schober Test will be performed. The examiner places the thumbs on the lower margin of the subject's upper posterior spines. An ink mark is drawn along the midline of the lumbar spine horizontal to the spines. While the examiner holds the tape measure firmly against the subject's skin, he or she marks a second line 15 cm above the original (upper mark). The subject is then asked to perform active anterior trunk flexion without increasing pain. The new distance between the lower and upper marks is measured. The subject returns to the neutral position. The difference in the initial distance between the marks in the neutral position and the new measurements taken in the flexion position is used to indicate the amount of lumbar flexion. After each measurement, the skin marks are removed with alcohol.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes